CLINICAL TRIAL: NCT00401141
Title: Phenotypic Characteristics and Transcriptomas of B Lymphocytes During Non Active Systemic Lupus Erythematosus
Brief Title: Abnormalities of B Lymphocytes During Systemic Lupus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 3156
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus; B lymphocytes; transcriptomas
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: Blood samples

SUMMARY:
Previous experimental data strongly suggest that B lymphocytes have intrinsic abnormalities during lupus in mice spontaneously affected by the disease. This study tries to define these abnormalities by looking at the gene expression profile of purified B lymphocytes from patients with non active systemic lupus , compared with the gene expression profile of purified B lymphocytes from healthy donnors.

ELIGIBILITY:
Inclusion criteria:

* non active systemic lupus

Exclusion criteria:

* immunosuppressive drugs
* more than 10 mg of prednisone per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pasquali, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service d'Immunologie Clinique et VIH - Hôpital Civil, Strasbourg, France

REFERENCES:
- [Result] Korganow AS, Knapp AM, Nehme-Schuster H, Soulas-Sprauel P, Poindron V, Pasquali JL, Martin T. Peripheral B cell abnormalities in patients with systemic lupus erythematosus in quiescent phase: decreased memory B cells and membrane CD19 expression. J Autoimmun. 2010 Jun;34(4):426-34. doi: 10.1016/j.jaut.2009.11.002. Epub 2009 Dec 5. PMID 19963348